CLINICAL TRIAL: NCT01584765
Title: Rechallenge Analysis: Detection of Potential Drug-Induced Liver Injury Using Kaiser California Database
Brief Title: Rechallenge, Potential Drug Induced Liver Injury (Kaiser)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115983; WEUKBRE5538 (Other: GSK)
Record Dates: First submitted 2012-04-12; First posted 2012-04-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Drug-induced Liver Injury
Keywords: liver injury; Rechallenge; Kaiser Permanente California
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Prescription Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Rechallenge: positive, negative, indeterminate and intermediate rechallenge subtypes
  Interventions: Drug: Prescription drugs with known hepatotoxicity
- Severe positive rechallenge: Subtype of positive rechallenge is defined as: ALT≥5 xULN or AP ≥2 xULN and bilirubin ≥2 xULN with one of the following: INR ≥1.5, Ascites, or Encephalopathy where time from liver chemistry elevation to INR≥1.5,ascites, or encephalopathy is less than 26 weeks in the absence of underlying cirrhosis; other organ failure considered due to DILI; liver-related hospitalization
  Interventions: Drug: Prescription drugs with known hepatotoxicity

INTERVENTIONS:
Drug: Prescription drugs with known hepatotoxicity — 14 prescription drugs with known hepatotoxicity : Amoxicillin/clavulanate, nitrofurantoin, isoniazid, trimethoprim-sulfamethoxazole, duloxetine, valproate, interferon-beta, ciprofloxacin, lamotrigine, phenytoin, diclofenac, terbinafine, levofloxacin, aripiprazole

SUMMARY:
Drug re-administration or rechallenge should be avoided after drug-induced liver injury (DILI) to avoid recurrent and fatal injury. Rechallenge outcomes vary considerably by drug and patient subjects. In order to better predict these outcomes, the objective of this analysis is to assess clinical outcomes of positive drug rechallenge following possible drug-induced liver injury. Electronic medical records from Kaiser Permanente California (KPSC), a managed care organization, will be utilized to identify patients who experience possible drug-induced liver injury following exposure to medications associated with hepatotoxicity, and who are then rechallenged with the medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received at least one prescription for a suspect drug between Jan 1, 2003 and June 30, 2009 (drug initiation period)
* Patients who experienced incident DILI event (identified by ALT ≥3xULN or AP ≥2xULN within 6 months of suspect drug administration) during the first exposure period that:

  1. Resolved to within normal limits of ALT (for hepatocellular & mixed) or AP (for cholestatic) within 180 days or
  2. Resolved to ALT < 3xULN (for hepatocellular & mixed) within 90 days or AP<2xULN (for cholestatic) within 180 days or
  3. Dropped by ≥50% of (Peak ALT - ULN) for hepatocellular or of (Peak AP - ULN) for cholestatic or mixed within 180 days
* Patients who were rechallenged with the same suspect drug; rechallenge will include first rechallenge event for the analysis.
* Patients who had at least of 12 months of continuous membership and drug benefit prior to and on the dispensing index date (inclusive). There is no minimum restriction of continuous membership plus drug benefit after the start date.
* Patients who were 18 years of age or older at the time of the first drug dispensing (index date) during the drug initiation period Jan 1, 2003 and June 30, 2009. Each patient's first prescription for the study drugs during the drug initiation period will be identified as index prescription.
* Patients who had health insurance coverage with full medical, pharmacy and lab benefits at the index date.

Exclusion Criteria:

* Patients meeting the definition of chronic liver injury and exhibiting persistent ALT≥3xULN or AP or bilirubin ≥2xULN within 90 days after initial injury
* Patients with chronic liver injury diagnostic codes or included in KPSC disease registries preceding the initial or rechallenge liver injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population was defined as patients 1) 18 years or older at the start of the drug exposure, 2) with 12 months or more of continuous membership plus drug benefit immediately prior to the drug start date, and 3) filling at least one prescription for fourteen drugs associated with hepatotoxicity (Chalasani 2008) anytime between Jan. 1, 2003 to June 30, 2009. Overall, 1,064,722 patients fulfill these criteria as derived from the total study population of the descriptive analysis. To be included in this analysis, patients had to be rechallenged with the same suspect drug and had at least one ALT measured at first exposure and during the rechallenge event. Study observations started in 2002 to allow for a year of pre-study observation in all exposures at risk. Applying all inclusion and exclusion criteria, the total study population comprises of 846 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Liver injury rechallenge | Up to seven and a half years
  Liver injury in relation to rechallenge types (positive, negative, indeterminate and intermediate) for hepatocellular, cholestatic and mixed DILI, respectively, defined according to Danan & Benichou, 1993, J Clin Epidemiol, 46(11): p. 1323-30.

SECONDARY OUTCOMES:
Severe positive rechallenge | Up to seven and a half years
  Severe positive rechallenge, defined as: ALT≥5 xULN or AP≥2 xULN and bilirubin≥2 xULN with one of the following: INR≥1.5, Ascites, or Encephalopathy where time from liver chemistry elevation to INR≥1.5,ascites, or encephalopathy<26 weeks in the absence of underlying cirrhosis; other organ failure considered due to DILI; or liver-related hospitalization. In subjects not meeting the definition of chronic liver injury and exhibiting persistent ALT≥3xULN or AP or bilirubin ≥2xULN after initial injury, positive drug rechallenge is defined as a doubling of ALT, alkaline phosphatase or bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline